CLINICAL TRIAL: NCT05179057
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial, With Cross-Over, of Posoleucel (ALVR105) for the Treatment of Adenovirus Infection in Pediatric and Adult Participants Receiving Standard of Care Following Allogeneic Hematopoietic Cell Transplantation
Brief Title: Posoleucel (ALVR105) for the Treatment of Adenovirus Infection in Pediatric and Adult Participants Receiving Standard of Care Following Allogeneic Hematopoietic Cell Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued as DSMB determined it was futile. No safety concerns were noted.
Sponsor: AlloVir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-105-303
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Adenovirus Infection
Keywords: Allogeneic Hematopoietic Cell Transplant; Adenoviremia; Adenovirus; Stem Cell Transplant; Posoleucel; ALVR105; Bone Marrow Transplant
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study with option for blinded crossover to assess the safety and efficacy of posoleucel as compared to placebo for the treatment of AdV infection in pediatric and adult recipients of HCT with AdV infections receiving SoC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Posoleucel + SoC (Experimental): Posoleucel + SOC; then placebo + SOC for patients who meet optional protocol-defined crossover criteria
  Interventions: Drug: Posoleucel
- Placebo + SoC (Placebo Comparator): Placebo + SOC; then Posoleucel + SOC for patients who meet optional protocol-defined crossover criteria
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Posoleucel — Administered as 2-4 milliliter infusion, visually identical to placebo
  Arms: Posoleucel + SoC
Drug: Placebo — Administered as 2-4 milliliter infusion, visually identical to Posoleucel
  Arms: Placebo + SoC

SUMMARY:
This study will assess the safety and efficacy of Posoleucel for the treatment of adenovirus (AdV) infection in pediatric and adult allo-HCT recipients receiving standard of care (SoC).

DETAILED DESCRIPTION:
During the period of immune recovery after allogeneic hematopoietic cell transplant (allo-HCT), viral infections and reactivations, including those with AdV, are an important cause of morbidity and mortality. Progression to AdV disease is associated with significant morbidity and mortality rates. This Phase 3, multicenter, randomized, double-blind, placebo-controlled study will assess the safety and efficacy of Posoleucel for the treatment of AdV infection in pediatric and adult allo-HCT recipients receiving SoC.

ELIGIBILITY:
Inclusion Criteria:

* Undergone allogeneic cell transplantation ≥21 days prior to dosing
* Meet one of the below criteria:

  1. AdV viremia DNA ≥10,000 copies/mL, OR
  2. AdV viremia DNA results of ≥1,000 copies/mL, AND

     1. has absolute lymphocyte count <180/mm3, OR
     2. has received T cell depletion OR
     3. had a cord blood transplant.

Exclusion Criteria:

* Grade 3 or higher acute GVHD
* Ongoing therapy with high-dose systemic corticosteroids
* Uncontrolled viral (other than AdV), bacterial, or fungal infection(s)
* Pregnant or lactating female unwilling to discontinue nursing prior to randomization
* History of severe prior reactions to blood product transfusions

NOTE: Other protocol-defined inclusion/exclusion criterion may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (23):
  - MD Anderson Cancer Center, Gilbert, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Lucile Packard Children's Hospital - Stanford University, Palo Alto, California
  - University of California, San Diego - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado - Center for Cancer and Blood Disorders, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida (UF) - Gainesville, Gainesville, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Texas Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Intermountain HealthCare - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Italy (8):
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - A.O.R.N. Santobono-Pausilipon, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Ospedale Regina Margherita, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale Borgo Trento, Verona
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital Lund, Lund
  - Karolinska University Hospital, Solna
- United Kingdom (8):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Children - Glasgow, Glasgow
  - University College London Hospital, London
  - St. Mary's Hospital, Paddington, London
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasileiou S, Kuvalekar M, Velazquez Y, Watanabe A, Leen AM, Gilmore SA. Phenotypic and functional characterization of posoleucel, a multivirus-specific T cell therapy for the treatment and prevention of viral infections in immunocompromised patients. Cytotherapy. 2024 Aug;26(8):869-877. doi: 10.1016/j.jcyt.2024.03.012. Epub 2024 Mar 19. PMID 38597860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 47 study centers in the United States, Canada, Italy, Spain, Sweden, and the United Kingdom, and participated from April 2022 to January 2024.
Pre-assignment Details: Participants with adenovirus infection receiving standard of care following allogeneic hematopoietic stem cell transplant (allo-HCT) were randomized in a 1:1 ratio to receive either posoleucel or placebo. Randomization was stratified by level of viremia (≥10,000 copies/mL or <10,000 copies/mL adenovirus DNA) and age (≥12 years or <12 years).
Groups:
- Posoleucel, Then Placebo: Participants were randomized to receive 2 sequential infusions of posoleucel, separated by 14 ± 3 days. The Primary Study Period included a 4-week efficacy evaluation followed by a 20-week safety follow-up.
  Eligible participants who experienced progression to active target organ disease or progression of existing target organ disease could cross-over to placebo treatment between Day 29 and Week 10. In the Cross-Over Period, participants received 2 sequential infusions of placebo, separated by 14 ± 3 days. The Cross-over Period included a 4-week efficacy evaluation followed by a 20-week safety follow-up.
- Placebo, Then Posoleucel: Participants were randomized to receive 2 sequential infusions of placebo, separated by 14 ± 3 days. The Primary Study Period included a 4-week efficacy evaluation followed by a 20-week safety follow-up.
  Eligible participants who experienced progression to active target organ disease or progression of existing target organ disease could cross-over to posoleucel treatment between Day 29 and Week 10. In the Cross-Over Period, participants received 2 sequential infusions of placebo, separated by 14 ± 3 days. The Cross-over Period included a 4-week efficacy evaluation followed by a 20-week safety follow-up.
Period: Overall Study
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Started | 30 | 27
Received Primary Study Treatment | 28 | 23
Met Cross-over Eligibility Criteria | 4 | 5
Received Cross-over Treatment | 4 | 5
Completed | 10 | 13
Not Completed | 20 | 14
Not completed — Adverse Event | 3 | 2
Not completed — Non-compliance with protocol requirements or study-related procedures | 1 | 0
Not completed — Study terminated | 13 | 7
Not completed — Discontinuation or withdrawal by participants/parent/legal guardian | 2 | 2
Not completed — Never received primary or cross-over study treatment | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (17.10) | 14.9 (15.80) | 15.6 (16.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 21 | 16 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5
  Black or African American | 3 | 1 | 4
  White | 19 | 20 | 39
  Not Reported | 3 | 1 | 4
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable Adenovirus Infection
Description: Viral load of adenovirus was measured at the central laboratory using quantitative polymerase chain reaction (qPCR) from blood and stool samples at each study visit and on Day 29 from a nasopharyngeal swab. There was a 14-day window for participants who crossed over from posoleucel to placebo; and for participants who crossed over from placebo to posoleucel, the pre-dose cross-over Day 1 viral load was used. Participants missing the primary endpoint but having undetectable viremia before Day 29 and after Day 43 were imputed as successes. Undetectable adenovirus viremia was less than the lower limit of quantification (LLOQ).
Time Frame: Day 29 through Day 43 (Day 29 + 14 days; up to 43 days post-first infusion)
Population: The modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of posoleucel or placebo. Only participants in the mITT population who completed through Day 29 or discontinued early were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Number analyzed (Participants) | 25 | 21
Participants | 11 | 9
Statistical Analysis 1: Comparison: Posoleucel, Then Placebo vs Placebo, Then Posoleucel; Test type: Superiority — A logistic regression model included treatment, level of viremia at baseline (≥10,000 copies/mL or <10,000 copies/mL adenovirus DNA), age (≥12 years or <12 years), and absolute lymphocyte counts at baseline. The null hypothesis is that the true percentage for posoleucel plus SoC is less than or equal to the true percentage for placebo plus SoC, and the alternative hypothesis is that it is greater; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.26 to 3.69] — Posoleucel versus Placebo

2. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) with a start date and time on or after the first dose of study treatment. A serious AE (SAE) was an AE that met at least one of the following serious criteria: fatal, life-threatening, required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; or other important medical event. TEAEs of special interest (AESI) included acute or chronic graft versus host disease, cytokine release syndrome, infusion-related reactions, and graft failure or rejection. Treatment-related refers to the assessment of a relationship between study treatment and the event by the investigator.
Time Frame: Up to 34 weeks
Population: The safety population included all participants who received any amount of posoleucel or placebo and had at least one post-treatment safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Posoleucel (Primary Study Period): Participants were randomized to receive 2 sequential infusions of posoleucel, separated by 14 ± 3 days, during the Primary Study Period.
- Placebo (Primary Study Period): Participants were randomized to receive 2 sequential infusions of placebo, separated by 14 ± 3 days, during the Primary Study Period.
- Posoleucel (Cross-over Period): Participants were randomized to receive 2 sequential infusions of placebo in the Primary Study Period and were eligible to cross-over between Day 29 and Week 10. Participants received posoleucel during the Cross-over Period.
- Placebo (Cross-over Period): Participants were randomized to receive 2 sequential infusions of posoleucel in the Primary Study Period and were eligible to cross-over between Day 29 and Week 10. Participants received placebo during the Cross-over Period.
Arm/Group | Posoleucel (Primary Study Period) | Placebo (Primary Study Period) | Posoleucel (Cross-over Period) | Placebo (Cross-over Period)
Number analyzed (Participants) | 28 | 23 | 5 | 4
Participants
  Any TEAE | 27 | 23 | 5 | 3
  Any TEAE related to study treatment | 7 | 9 | 1 | 1
  Any AESI | 6 | 9 | 1 | 2
  Any SAE | 16 | 16 | 3 | 1
  Any SAE related to study treatment | 1 | 1 | 1 | 1
  Any TEAE leading to study treatment discontinuation | 2 | 1 | 0 | 2
  Any TEAE leading to study discontinuation | 1 | 2 | 0 | 1
  Any TEAE leading to death | 2 | 1 | 0 | 1

3. Secondary Outcome: Number of Participants With Overall Disease Progression
Time Frame: From Day 29 up to Week 10
Population: Data not collected due to early termination after Data and Safety Monitoring Board (DSMB) futility analysis concluded the study was unlikely to meet its primary endpoint.
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Area Under the Curve (AUC) Adenovirus Viral Load
Time Frame: Pre-dose and Day 29
Population: Data not collected due to early termination after DSMB futility analysis concluded the study was unlikely to meet its primary endpoint.
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Who Achieved Adenovirus Viremia <400 Copies/mL at Day 29
Time Frame: Day 29
Population: as for outcome 4
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Undetectable Adenovirus Viremia (Less Than LLOQ)
Time Frame: Pre-dose to 34 weeks
Population: as for outcome 4
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Adenovirus Disease Recurrence
Time Frame: 34 weeks
Population: as for outcome 4
Arm/Group | Posoleucel, Then Placebo | Placebo, Then Posoleucel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 34 weeks
Arm/Group | Posoleucel (Primary Study Period) | Placebo (Primary Study Period) | Posoleucel (Cross-over Period) | Placebo (Cross-over Period)
All-Cause Mortality (participants affected / at risk) | 2/28 | 1/23 | 0/5 | 1/4
Serious Adverse Events (participants affected / at risk) | 16/28 | 16/23 | 3/5 | 1/4
Other Adverse Events (participants affected / at risk) | 27/28 | 23/23 | 5/5 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (Primary Study Period) (N=28) | Placebo (Primary Study Period) (N=23) | Posoleucel (Cross-over Period) (N=5) | Placebo (Cross-over Period) (N=4)
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Cryptosporidiosis infection (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Pancreatitis viral (Infections and infestations) | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Phlebitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 3 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chronic graft versus host disease in intestine (Immune system disorders) | 1 | 1 | 0 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 0 | 0 | 0
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1 | 0 | 0
Chronic graft versus host disease (Immune system disorders) | 0 | 1 | 0 | 0
Chronic graft versus host disease in lung (Immune system disorders) | 0 | 1 | 0 | 0
Chronic graft versus host disease oral (Immune system disorders) | 1 | 0 | 0 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 1 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Immune-mediated cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal tubular disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (Primary Study Period) (N=28) | Placebo (Primary Study Period) (N=23) | Posoleucel (Cross-over Period) (N=5) | Placebo (Cross-over Period) (N=4)
COVID-19 (Infections and infestations) | 3 | 1 | 0 | 1
Rhinovirus infection (Infections and infestations) | 2 | 3 | 0 | 0
BK virus infection (Infections and infestations) | 3 | 1 | 0 | 0
Candida infection (Infections and infestations) | 2 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 3 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 3 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 3 | 0 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 1 | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Adenoviral hepatitis (Infections and infestations) | 2 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 2 | 0 | 0 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 | 1 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 2 | 0 | 0 | 0
Epstein-Barr viraemia (Infections and infestations) | 1 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 1 | 0
Viral rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 3 | 1 | 0
Weight decreased (Investigations) | 2 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 2 | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 1
Enterobacter test positive (Investigations) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 6 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
Pyrexia (General disorders) | 10 | 8 | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 5 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 3 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 3 | 0 | 0
Acute graft versus host disease in skin (Immune system disorders) | 2 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 3 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1
Graft versus host disease in liver (Immune system disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 1 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 4 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0
Orbital haematoma (Eye disorders) | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued following a pre-planned DSMB futility analysis concluding that the study was unlikely to meet its primary endpoint, no safety concerns were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT05179057/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT05179057/SAP_001.pdf